CLINICAL TRIAL: NCT05959577
Title: A Randomized Prospective Clinical Trial Comparing the Surgical Outcomes of Traditional Ferguson Hemorrhoidectomy Versus Stapled Hemorrhoidopexy With Anoplasty for Patients With Grade III/IV Hemorrhoids
Brief Title: Traditional Ferguson Hemorrhoidectomy vs Stapled Hemorrhoidopexy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207069RINB
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Haemorrhoid
Keywords: Hemorrhoid; Ferguson hemorrhoidectomy; Stapled hemorrhoidopexy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferguson hemorrhoidectomy (Experimental): The patients who meet the inclusion and exclusion criteria in this group will undergo Ferguson hemorrhoidectomy
  Interventions: Procedure: Ferguson hemorrhoidectomy
- Stapled hemorrhoidopexy with anoplasty (Active Comparator): The patients who meet the inclusion and exclusion criteria in this group will undergo Stapled hemorrhoidopexy with anoplasty
  Interventions: Procedure: Stapled hemorrhoidopexy with anoplasty

INTERVENTIONS:
Procedure: Stapled hemorrhoidopexy with anoplasty — The patients who meet the inclusion and exclusion criteria in this group will undergo Stapled hemorrhoidopexy with anoplasty.
  Arms: Stapled hemorrhoidopexy with anoplasty
Procedure: Ferguson hemorrhoidectomy — Ferguson hemorrhoidectomy
  Arms: Ferguson hemorrhoidectomy

SUMMARY:
This study aimed to compare the short- and long-term outcomes of stapled hemorrhoidopexy (the procedure for prolapsed hemorrhoids, PPH) with anoplasty versus traditional Ferguson method for the treatment of patients with grade III /IV hemorrhoids.

DETAILED DESCRIPTION:
Hemorrhoidal disease is a common pathology affecting 5 percent of the general population. Hemorrhoidectomy is the most effective approach for hemorrhoidal disease, especially for Grade III and IV hemorrhoids, and is one of the most frequently performed general surgeries. For patients with circumferential prolapsed hemorrhoids, the standard three-quadrant hemorrhoidectomy (Milligan-Morgan or Ferguson method) may leave behind too much hemorrhoid-bearing mucosa and skin tags, which are the main complaints of patients as incomplete resection or recurrence. Since its first description in 1882, the Whitehead hemorrhoidectomy has earned a reputation as a radical procedure for circumferential prolapsed hemorrhoids. However, this procedure has been criticized because it is time-consuming and causes considerable blood loss, disturbed continence, ectropion of the rectal mucosa, and stricture formation, and it has been used rarely by surgeons. More recent modifications, such as a circular incision, anodermal flap graft, or sliding skin flap graft, reduce the risk of complications associated with the primary method, but the results remain unsatisfactory. Some colorectal surgeons have used a modified Ferguson method with various degrees of anoplasty and an anodermal flap to treat circumferential hemorrhoids during the past 20 years,8 but unsatisfactory results were still experienced, including occasional flap necrosis, which causes skin defects and anal stenosis. Furthermore, the loss of most cushioning effect of the anus, which results in varying degrees of incontinence, also is a problem. Stapled hemorrhoidopexy was presented as a procedure for prolapsed hemorrhoids (PPH) in 1998 by Longo. From the viewpoints of lesser post operative pain and short recuperation period after PPH, it was later adapted for grade III and grade IV hemorrhoids gradually. However, PPH had several drawbacks and long-term sequelae, such as residual skin tags, anal stenosis and even chronic anal pain after surgery. Therefore, the Milligan- Morgan hemorrhoidectomy (MMH) or modified Ferguson method is still the most popular method for hemorrhoids. The explanation for residual skin tags is probably that the external components remained untreated by stapling in most of the studies. Therefore, we have been routinely adding an anoplasty for the prominent skin tag after the stapling hemorrhoidopexy procedure. Moreover, previous studies have demonstrated a reduction of rectal distensibility and volume thresholds for sensations in patients treated with stapled hemorrhoidopexy, and a possible correlation between rectal functional alterations and postoperative disorders was postulated. The present study aimed to compare the short- and long-term outcomes of PPH with anoplasty and traditional Ferguson hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25~75 years with subjective, severe hemorrhoidal symptoms
* Graded III-IV hemorrhoid
* The patients' condition can undergo hemorrhoidectomy
* ASA status ≤ 3

Exclusion Criteria:

* Severe liver cirrhosis
* Chronic renal disease
* Coagulopathy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 6 months
  Recorded with visual analogue scale (VAS)

SECONDARY OUTCOMES:
Time to normal life or work | 6 months
  The recovery duration before the patient returns to their normal life
Post-operative anal hemorrhage | 6 months
  Any bleeding needs medicines or surgical intervention
Wound dehiscence or discharge | 6 months
  Diagnosed as the presence of open wound needs oral or intravenous antibiotics treatment or surgical dressing
Pruritus | 6 months
  The presence of pruritus that needs topical ointment or antihistamine to relieve the symptom
Urinary retention | 6 months
  No urination for four hours; urinary retention within bladder > (body weight ) x 4 hours confirmed by ultrasound; the patient needs catheterization.
Sphincter damage | 6 months
  Measured by digital examination

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, MD, Study Director — National Taiwan University Hospital
Locations (1):
- Jin-Tung LIANG, Taipei, Taiwan